CLINICAL TRIAL: NCT05247021
Title: Bilateral Ultrasound Guided Erector Spinae Plane Block for Postoperative Pain Management in Lumbar Spine Surgery ( a Controlled Study Trial)
Brief Title: Erector Spinae Plane Block in Spine Surgeries
Acronym: ESB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ainshmas university
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Lumbar Disc Disease
Keywords: erector spinae block; Lumbar disc surgery
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae block group (E) (Experimental): patients will receive bilateral ultrasound guided erector spinae block before the lumbar spine surgery starts.(20ml of bupivacaine 0.25%) after receiving general anesthesia
  Interventions: Procedure: erector spinae block for group E
- control group (C) (No Intervention): patients will receive standard general anesthesia for lumbar spine surgery according to hospital protocol.

INTERVENTIONS:
Procedure: erector spinae block for group E — . The patient will be placed in the prone position. A high-frequency linear probe or a curved array probe, depending on the BMI of the patient, will be placed in longitudinal alignment, 2-3cm lateral to the vertebral column. The transverse processes of the vertebrae at the level of surgery, the erector spinae muscle, and the psoas muscle will be identified. A 5- or 8-cm 22-G ultrasound needle will be inserted with an in-plane technique in a cephalad-to-caudal direction until bone contact with the top of the transverse process is reached. After slight retraction of the needle, 20ml of bupivacaine 0.25% will be injected behind the erector spinae muscle. The same procedure will be repeated on the contralateral side.
  Arms: erector spinae block group (E)

SUMMARY:
Aim of this study was to assess the efficacy of erector spinae plane block (ESB) for postoperative pain management in lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anesthesiologists physical status (ASA) I and II.
* Both sexes.
* Age between 20 to 60 years old.
* Scheduled for lumbar spine surgeries.

Exclusion Criteria:

* Patients who received long acting opioids preoperatively.
* Patients with bleeding disorders and coagulopathy.
* Infection at the injection site.
* Allergy to local anesthetics.
* Patients with significant cognitive dysfunction.
* Patients with diabetic neuropathy.
* Patients with uncontrolled hypertension or diabetes.
* Patients with advanced cardiac, respiratory, hepatic or renal disease.
* Patients with viral hepatitis or HIV.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
the postoperative 24 hours morphine consumption | 24 hours postoperative
  the analgesic effect of erector spine block will be assessed postoperative by numeric rating scale (NRS), if NRS is more than 3 the patient will receive a rescue dose of 5 milligrams of morphine

SECONDARY OUTCOMES:
Mean Blood pressure in mmHg | 24 hours postoperative
  Measure mean blood pressure of patients postoperative every 4 hours
Heart rate | 24 hours postoperative
  Measure heart of the patients postoperative every 4 hours
Patient satisfaction | 24 hours postoperative
  Measure patient satisfaction by asking the patient if he is satisfied or not " yes or no"
First time of mobilization to a chair | 24 hours postoperative
  Measure the time to first mobilization to a chair in minutes

CONTACTS AND LOCATIONS:
Overall Officials: ossama mansour, professor, Study Chair — faculty of medicine , ain shams university
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625